CLINICAL TRIAL: NCT06630702
Title: Application of Thoracic Epidural Spinal Cord Stimulation (SCS) for Managing Freezing of Gait (FOG) in Patients With Advanced Parkinson's Disease
Brief Title: Application of Thoracic Epidural SCS for Managing FOG in Patients With Advanced Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202307093DINC
Record Dates: First submitted 2024-09-18; First posted 2024-10-08 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Parkinson Disease; Freezing of Gait; Spinal Cord Stimulation
Keywords: Spinal cord stimulation, Freezing of gait; Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- SCS implantation (Experimental)
  Interventions: Device: SCS electrode stimulation 1; Device: SCS electrode stimulation 2; Device: SCS electrode stimulation 3

INTERVENTIONS:
Device: SCS electrode stimulation 1 — 300Hz/300us
Device: SCS electrode stimulation 2 — 130Hz/300us
Device: SCS electrode stimulation 3 — 60Hz/300us

SUMMARY:
Spinal cord stimulation (SCS) has proven to be effective for pain that is unresponsive to medication. This technique involves an anesthesiologist or a neurosurgeon placing stimulation electrodes at the thoracic vertebrae to provide pain relief. Although SCS is not currently a standard treatment for patients with Parkinson's disease, recent studies have shown that Parkinson's patients who experience intolerable pain and undergo SCS treatment not only experience pain relief but also show improvements in gait and other Parkinson's symptoms. Therefore, the investigators aim to use temporary, minimally invasive SCS electrodes to help patients with nrFOG (non-responsive Freezing of Gait) improve their stability and reduce their risk of falls.

ELIGIBILITY:
Inclusion Criteria:

* Age:40-85 years old.
* Patients with primary Parkinson's disease who have been diagnosed by a movement disorder specialist for more than 5 years. Although they have a clear response to drugs, they have a frozen gait that cannot be controlled by drugs. Lower limb pain may be present with or without Parkinson's non-motor symptoms.
* No other secondary gait problems.

Exclusion Criteria:

* Atypical Parkinson's disease.
* Patients with spinal cord injuries.
* Medication-controlled frozen gait.
* It is expected that there are lesions near the implantation area causing spinal canal stenosis or myelopathy (can be ruled out by MRI).
* It is expected that the implantation area has undergone previous surgery or there is infection near the implantation area, which may affect the success rate of implantation or increase concerns about complications (such as severe extraspinal adhesion, or spinal cord damage in previous surgeries).
* People with abnormal coagulation function (such as hemophilia patients) or those who have been controlled by long-term use of antithrombotic drugs and cannot stop taking them in a short period of time.
* CDR (Clinical Dementia Rating Scale) ≧2. 8. Those who are allergic to developer.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Gait parameters --- foot rotation [degtree] | Day 0, Day 2, Day 3, Day 4, and Day 7
  (1)Measured by plantar pressure distribution measurement systems (100 Hz, FDM-T, Zebris Medical GmbH, Germany) with a maximum gait track of 6 meters.
Gait parameters --- step length [cm] | Day 0, Day 2, Day 3, Day 4, and Day 7
  (1)Measured by plantar pressure distribution measurement systems (100 Hz, FDM-T, Zebris Medical GmbH, Germany) with a maximum gait track of 6 meters.
Gait parameters --- stride length [cm] | Day 0, Day 2, Day 3, Day 4, and Day 7
  (1)Measured by plantar pressure distribution measurement systems (100 Hz, FDM-T, Zebris Medical GmbH, Germany) with a maximum gait track of 6 meters.
Gait parameters --- step width [cm] | Day 0, Day 2, Day 3, Day 4, and Day 7
  (1)Measured by plantar pressure distribution measurement systems (100 Hz, FDM-T, Zebris Medical GmbH, Germany) with a maximum gait track of 6 meters.
Gait parameters --- stance phase [%] | Day 0, Day 2, Day 3, Day 4, and Day 7
  (1)Measured by plantar pressure distribution measurement systems (100 Hz, FDM-T, Zebris Medical GmbH, Germany) with a maximum gait track of 6 meters.
Gait parameters --- swing phase [%] | Day 0, Day 2, Day 3, Day 4, and Day 7
  (1)Measured by plantar pressure distribution measurement systems (100 Hz, FDM-T, Zebris Medical GmbH, Germany) with a maximum gait track of 6 meters.
Gait parameters --- double stance phase [%] | Day 0, Day 2, Day 3, Day 4, and Day 7
  (1)Measured by plantar pressure distribution measurement systems (100 Hz, FDM-T, Zebris Medical GmbH, Germany) with a maximum gait track of 6 meters.
Gait parameters --- step time [second] | Day 0, Day 2, Day 3, Day 4, and Day 7
  (1)Measured by plantar pressure distribution measurement systems (100 Hz, FDM-T, Zebris Medical GmbH, Germany) with a maximum gait track of 6 meters.
Gait parameters --- stride time [second] | Day 0, Day 2, Day 3, Day 4, and Day 7
  (1)Measured by plantar pressure distribution measurement systems (100 Hz, FDM-T, Zebris Medical GmbH, Germany) with a maximum gait track of 6 meters.
Gait parameters --- cadence [steps/minute] | Day 0, Day 2, Day 3, Day 4, and Day 7
  (1)Measured by plantar pressure distribution measurement systems (100 Hz, FDM-T, Zebris Medical GmbH, Germany) with a maximum gait track of 6 meters.
Gait parameters --- velocity [km/hour] | Day 0, Day 2, Day 3, Day 4, and Day 7
  (1)Measured by plantar pressure distribution measurement systems (100 Hz, FDM-T, Zebris Medical GmbH, Germany) with a maximum gait track of 6 meters.

SECONDARY OUTCOMES:
Clinical Scale | Day 0, Day 2, Day 3, Day 4, and Day 7
  1. Tinetti Gait Analysis
  2. Score: 0-16 (Higher scores means better.)
Clinical score | Day 0, Day 2, Day 3, Day 4, and Day 7
  1. MDS-UPDRS part III (motor examination)
  2. Score: 0-72 (Higher scores means worse.)
Clinical Scale | Day 0, Day 2, Day 3, Day 4, and Day 7
  1. Time up and Go test
  2. Patients wear their regular footwear and can use a walking aid, if needed. Begin by having the patient sit back in a standard arm chair and identify a line 3 meters, or 10 feet away, on the floor.
  3. Score: Time in Seconds (Shorter time means better.)
Clinical Scale | Day 0, Day 2, Day 3, Day 4, and Day 7
  1. Freezing of gait questionnaire
  2. Score: 0-26 (Higher scores means worse.)
Clinical Scale | Day 0, Day 2, Day 3, Day 4, and Day 7
  1. Activities-specific balance confidence scale
  2. Score:0%-100% (Higher percentage means better.)

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital Hsin-Chu Branch, Hsinchu, Hsinchu City, Taiwan